CLINICAL TRIAL: NCT03718247
Title: The Effect of the Ketogenic Diet on Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Utilization of the Ketogenic Diet in Patient With Relapsing Remitting MS
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, J. Nicholas Brenton, MD, Assistant Professor of Neurology and Pediatrics, University of Virginia
Other Study IDs: 20877
Record Dates: First submitted 2018-10-16; First posted 2018-10-24 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Ketogenic diet
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Rectal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Modified Atkins diet — High fat low carbohydrate diet.

SUMMARY:
The purpose of this study is to evaluate the benefits of a low-carbohydrate, high-fat diet (ketogenic diet) in up to 50 subjects with relapsing-remitting multiple sclerosis (RRMS), a chronic neuro-inflammatory disease. The primary aim of this study is to provide evidence of tolerability of the ketogenic diet in patients with RRMS. The principal investigator hypothesizes that the diet may prove beneficial for participants disease state in multiple potential ways.The study consists of 5 visits over a 12 month period. During these visits subjects will undergo fasting lab work, micro-biome sampling, neurological testing, body composition analysis, meeting with dietitian, and will be asked to complete surveys as well as a diet recall log.

DETAILED DESCRIPTION:
The purpose of this study is to see if a high fat, low carbohydrate diet is safe and how it effects post trial diet habits, physique, and disease course in patients with relapsing remitting multiple sclerosis. In particular, multiple sclerosis is a neurodegenerative disorder that is characterized by inflammation, microglial inflammation, and hypoxia in its relapsing-remitting form.1 One of the hypothesized therapeutic mechanisms of ketogenic diets is related to its effect on decreasing glycolysis, decreasing reactive oxygen species (ROS), and increasing ATP production by mitochondria. Production of ROS and macrophage activation have been directly correlated with demyelination and axonal injury in multiple sclerosis.2,3 In mouse models with experimental allergic encephalomyelitis (EAE), a model disease in mice that has many similar properties to that of MS in humans, experiments have demonstrated that impairment of memory and spatial learning are directly correlated with increased cytokine and chemokine expression and ROS production. In EAE mice fed a ketogenic diet, there were noted improvements in motor disability, memory dysfunction, and CNS inflammation - which on the whole are suggestive that a ketogenic diet may have a multitude of benefits in patients with multiple sclerosis.

The study goal is to recruit 50 young adult or adult patients with relapsing-remitting multiple sclerosis that show interest in starting and maintaining a ketogenic diet for six months. Prior to initiating the diet, the study team will characterize each patient's disease by analyzing multiple factors - including baseline expanded disability status scale (EDSS) and annualized relapse rates (ARR). Throughout the course of the 12 month study participants will be asked to complete several patient reported outcomes, an online food diary recall, and track their diet compliance using urinary ketone testing strips provided by the study daily.In addition, the study team will also draw serum lab work every 3 months that we anticipate may be affected by the diet (including hemoglobin A1C, lipid panel, and cytokine profiles). Rectal swabs will be requested during the study to look at effects of the diet on the microbiome both pre and post diet. Additionally, activity monitors (accelerometers) will be worn by each subject for 1 week prior to initiation of the diet to provide evidence of pre-diet activity levels and at various times throughout the study for comparison. Participating patients will receive education on starting, maintaining, and stopping the 6 month diet by a nutritionist. The nutritionist will meet with patients at scheduled office visits and will be available for questions during the duration of the patients participation. Subjects will also undergo anthropometric assessments with a bodpod used to measure body mass as well.

All measures will be compared with statistical analyses, utilizing both pre and post diet values to help determine benefit of the diet on various aspects of the patient's overall health and wellness.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent (or assent for minors)
2. Relapsing-remitting MS diagnosis per 2010 McDonald criteria
3. On same Demyelinating Treatment for at least 6 months
4. Ages ≥ 12 years to ≤ 45 years

Exclusion Criteria:

1. Comorbid disease (including hypercholesterolemia, cardiovascular or renal disease) that would interfere with safety and/or study completion
2. Current pregnancy or planning pregnancy
3. Progressive form of MS
4. Estimated GFR less than 45 mL/min based on a serum creatinine drawn within 30 days of enrollment
5. Acute kidney injury
6. History of paraproteinemia syndromes such as multiple myeloma
7. Hepatorenal syndrome
8. Liver transplant
9. Underweight or low weight patients as defined by:

   1. BMI value <20 for those 18 years and older
   2. <10th percentile for BMI by CDC growth charts for those less than 18 years of age

Ages: 12 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with relapsing-remitting MS
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-10-31 (Actual); Primary Completion 2021-06-21 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Diet Tolerability and compliance | 6 months
  Determine if patients are able to adhere to (number of days patient able to demonstrate ketosis) and tolerate a strict diet over an extended period of time as reported in urinary ketone analysis.
Diet Benefits | 12 months
  Determine the benefits, if any, of the ketogenic diet in RRMS subjects physically, emotionally, and clinically as reported in patient reported outcome surveys. Survey responses are evaluated on a scale of 0-10 with 0 being no affect and 10 being highly affected by the disease.

SECONDARY OUTCOMES:
Physical changes | 12 months
  Assessment of height and weight to calculate subject BMI throughout the study. This will be compared with survey on physical activity to see if scores (no disease impact to high disease impact on activity) correspond with changes in BMI.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

REFERENCES:
- [Background] Zhao Z, Lange DJ, Voustianiouk A, MacGrogan D, Ho L, Suh J, Humala N, Thiyagarajan M, Wang J, Pasinetti GM. A ketogenic diet as a potential novel therapeutic intervention in amyotrophic lateral sclerosis. BMC Neurosci. 2006 Apr 3;7:29. doi: 10.1186/1471-2202-7-29. PMID 16584562
- [Background] Lassmann H, van Horssen J, Mahad D. Progressive multiple sclerosis: pathology and pathogenesis. Nat Rev Neurol. 2012 Nov 5;8(11):647-56. doi: 10.1038/nrneurol.2012.168. Epub 2012 Sep 25. PMID 23007702
- [Background] van Horssen J, Schreibelt G, Drexhage J, Hazes T, Dijkstra CD, van der Valk P, de Vries HE. Severe oxidative damage in multiple sclerosis lesions coincides with enhanced antioxidant enzyme expression. Free Radic Biol Med. 2008 Dec 15;45(12):1729-37. doi: 10.1016/j.freeradbiomed.2008.09.023. Epub 2008 Oct 7. PMID 18930811
- [Derived] Perlman J, Wetmore E, Lehner-Gulotta D, Banwell B, Bergqvist AGC, Coleman R, Chen S, Conaway M, Goldman MD, Morse AM, Brenton JN. Impact of a ketogenic diet on sleep quality in people with relapsing multiple sclerosis. Sleep Med. 2024 Oct;122:213-220. doi: 10.1016/j.sleep.2024.08.020. Epub 2024 Aug 28. PMID 39208520
- [Derived] Wetmore E, Lehner-Gulotta D, Florenzo B, Banwell B, Bergqvist AGC, Coleman R, Conaway M, Goldman MD, Brenton JN. Ketogenic diet in relapsing multiple sclerosis: Patient perceptions, post-trial diet adherence & outcomes. Clin Nutr. 2023 Aug;42(8):1427-1435. doi: 10.1016/j.clnu.2023.06.029. Epub 2023 Jul 4. PMID 37433230
- [Derived] Oh U, Woolbright E, Lehner-Gulotta D, Coleman R, Conaway M, Goldman MD, Brenton JN. Serum neurofilament light chain in relapsing multiple sclerosis patients on a ketogenic diet. Mult Scler Relat Disord. 2023 May;73:104670. doi: 10.1016/j.msard.2023.104670. Epub 2023 Mar 25. PMID 36996634
- [Derived] Brenton JN, Lehner-Gulotta D, Woolbright E, Banwell B, Bergqvist AGC, Chen S, Coleman R, Conaway M, Goldman MD. Phase II study of ketogenic diets in relapsing multiple sclerosis: safety, tolerability and potential clinical benefits. J Neurol Neurosurg Psychiatry. 2022 Jun;93(6):637-644. doi: 10.1136/jnnp-2022-329074. Epub 2022 Apr 13. PMID 35418509